CLINICAL TRIAL: NCT05926778
Title: Multiomics Study of Fibrosis Factors After Liver Transplantation and Exploration of Fibrosis Methylation Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Renji-LY2023-075-B
Record Dates: First submitted 2023-06-06; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Liver Fibrosis
Keywords: Liver Fibrosis; Liver Transplantation; Biomarkers; DNA methylation
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood and liver puncture biopsy specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibrosis Cohort: Adult(10 patients) and pediatric(10 patients) liver transplant recipients with fibrosis determined by histological examination of liver biopsy
  Interventions: Other: Liver allograft fibrosis
- Control Cohort: Adult(20 patients) and pediatric(20 patients) liver transplant recipients without fibrosis determined by histological examination of liver biopsy

INTERVENTIONS:
Other: Liver allograft fibrosis — Observational studies without intervention
  Groups: Fibrosis Cohort

SUMMARY:
This is a retrospective observational study in liver transplantation recipients with or without allograft liver fibrosis. Based on the GM-seq and Tcr-Seq data, a novel diagnostic model including DNA-methylation and TCR-Seq biomarkers will be established.

DETAILED DESCRIPTION:
This is a retrospective study on 60 patients who had previously received liver transplantation in our hospital. The patients will be stratified according to age, including 20 children and 20 adults with allograft liver fibrosis after liver transplantation, while 10 children and 10 adults with fibrosis, respectively.

1. The differential analysis of DNA-methylation will be performed between the allograft liver fibrosis cohort and the control cohort based on the GM-seq sequencing data. And the fibrosis-specific DNA-methylation CpG sites or regions in liver and peripheral blood will be explored in the liver transplantation recipients.
2. The abundance and diversity of TCR between the allograft liver fibrosis cohort and the control cohort will be analyzed. And the fibrosis-specific TCR sequence of allograft liver fibrosis will be screened based on TCR-Seq sequencing and tNGS.
3. The characteristics of DNA-methylation and TCR-Seq biomarkers in allograft liver fibrosis population will be defined. And the similarities and differences of the characteristics between children and adults will be explored.
4. Based on the GM-seq and Tcr-Seq data, a novel diagnostic model including DNA-methylation and TCR-Seq biomarkers will be established.

ELIGIBILITY:
Inclusion Criteria:

1. Living donor liver transplantation of left outer lobe or left half liver for biliary atresia in children (≤18 years old), or orthotopic liver transplantation for hepatitis B cirrhosis in adults (> 18 years old), regardless of gender;
2. Oral tacrolimus immunosuppressive therapy;
3. Received liver transplantation in our hospital for the first time and did not receive liver transplantation again;
4. Patients need to be admitted to hospital for programmed liver biopsy or receive liver biopsy due to abnormal liver function;
5. Complete clinical data and samples (including liver puncture biopsy specimens, plasma, and PBMC of the same period);
6. The subjects or their guardians voluntarily join the study, sign the informed consent, comply well, and cooperate with follow-up.

Exclusion Criteria:

1. Combined multi-organ transplantation;
2. Pregnancy or lactation;
3. Severe systemic infection;
4. Contraindications of liver biopsy with multiple organ failure or coagulation dysfunction;
5. Previous history of allergy to narcotic or sedative drugs;
6. In the stage of acute rejection hormone shock therapy;
7. Incomplete clinical data and samples;
8. Situations considered unsuitable for inclusion by other researchers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult or pediatric recipients who underwent liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensivity | 7 Days
  Sensivity is the true positive rate of the novel diagnostic model [Liver fibrosis is determined by histological examination of liver biopsy (LAFSc)].
Specificity | 7 Days
  Specificity is the true negative rate of the novel diagnostic model [Liver fibrosis is determined by histological examination of liver biopsy (LAFSc)].
AUROC | 7 Days
  AUROC is the area under the receiver operating characteristic curve [Liver fibrosis is determined by histological examination of liver biopsy (LAFSc)].

SECONDARY OUTCOMES:
Heterogeneity of the DNA-methylation biomarkers in allograft liver fibrosis cohort | 7 Days
  The similarities and differences of the characteristics of DNA-methylation and TCR-Seq biomarkers between children and adults in the allograft liver fibrosis cohort.
Heterogeneity of the TCR-Seq biomarkers in allograft liver fibrosis cohort | 7 Days
  The similarities and differences of the characteristics of TCR-Seq biomarkers between children and adults in the allograft liver fibrosis cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, Prof. MD, Study Chair — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU; Hao Feng, MD., Ph.D., Principal Investigator — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No